CLINICAL TRIAL: NCT03161964
Title: Propranolol as a Treatment for Impaired Awareness of Hypoglycemia in Type 1 Diabetes
Brief Title: Propranolol in Treating Hypoglycemia Unawareness
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Statistical power could not be achieved due to low enrollment.
Sponsor: Anu Sharma (Other)
Responsible Party: Sponsor-Investigator, Anu Sharma, Principal Investigator; Assistant Professor (Clinical), University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB #101995
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Hypoglycemia; Impaired Awareness of Hypoglycemia; Propranolol
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Propranolol; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): After enrollment and the initial two-week continuous glucose monitoring assessment, study subjects randomized to the Propranolol Arm will be treated with Propranolol 80 Mg Oral Capsule, Extended Release daily for four weeks.
  Interventions: Drug: Propranolol 80 Mg Oral Capsule, Extended Release
- Placebo (Experimental): After enrollment and the initial two-week continuous glucose monitoring assessment, study subjects randomized to the Placebo Arm will be treated with matching placebo oral capsule daily for four weeks.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Propranolol 80 Mg Oral Capsule, Extended Release — Propranolol capsule over-encapsulated to match placebo for blinding
  Other Names: propranolol Long Acting (LA)
  Arms: Propranolol
Drug: Placebo oral capsule — Placebo capsule over-encapsulated to match propranolol for blinding
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Impaired awareness of hypoglycemia is common in type 1 diabetes (T1DM) patients. Impaired hypoglycemia awareness increases severe hypoglycemia risk by six-fold. Severe hypoglycemia compromises quality of life and can potentially cause death. The long-term goal of this pilot study is to lead to the development of novel therapeutic approaches to improve hypoglycemia awareness and thus prevent severe hypoglycemia development in T1DM population with impaired awareness of hypoglycemia.

It is hypothesized that propranolol will improve hypoglycemia recognition in T1DM. The specific aims of the study are to determine whether propranolol treatment improves subjects' recognition of hypoglycemic episodes, and improves hypoglycemic awareness scores; whether propranolol favorably increases hypoglycemia blood glucose nadir, decreases onset-to-treatment/recovery time (i.e. hypoglycemia duration), and reduces hypoglycemia/severe hypoglycemia frequency; and, whether propranolol reduces fear of hypoglycemia and improves overall blood glucose control.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) can lead to serious and devastating complications, including microvascular (retinopathy, neuropathy and nephropathy) and cardiovascular disease. Both diabetic microvascular and cardiovascular complications can be reduced with intensive insulin therapy and strict blood glucose control which target hemoglobin A1C to less than 7%. However, tighter glycemic control correlates with a higher incidence of hypoglycemia and severe hypoglycemia. Recurring exposure to hypoglycemia leads to an attenuated sympathoadrenal response to hypoglycemia (which is termed hypoglycemia-associated autonomic failure), and thus a loss or decrease in neurogenic hypoglycemic symptoms (i.e. impaired awareness of hypoglycemia). Impaired awareness of hypoglycemia is associated with a six-fold increased risk of severe hypoglycemia and physician or patient-directed higher glycemic goals. Impaired awareness of hypoglycemia is therefore a major barrier in diabetes management, by precluding optimal glycemic control and realization of its full benefits.

Several therapeutic strategies have been proposed to improve hypoglycemia awareness in T1DM patients. A temporal increase in glycemic goal only sustains hypoglycemia awareness recovery for a short-term. Islet transplantation is invasive, extremely expensive and requires life-long use of immunosuppressants. A widely available and affordable treatment with sustained efficacy for improving hypoglycemia awareness is therefore in urgent need. Pharmaceutical agents targeting potential mechanisms that contribute to the development of impaired hypoglycemia awareness have been proposed, including beta-blockers, opioid receptor antagonists and selective serotonin uptake inhibitors (SSRIs). However, none of these agents has been approved for the treatment of impaired hypoglycemia awareness.

The current pilot study will examine the clinical use of beta-blockers, specifically propranolol, for the treatment of impaired hypoglycemia awareness. In a physiological condition, hypoglycemia leads to counterregulatory hormone responses, including catecholamines. Catecholamine elevation mediates the development of neurogenic symptoms, including palpitation, anxiety and diaphoresis, and patient's recognition of a hypoglycemic episode. Previous study suggests that recurring hypoglycemic events, potentially through repeated ventromedial hypothalamus (VMH) noradrenergic system activation, dampen the counterregulatory hormone response to hypoglycemia. In addition, carvedilol (a non-specific beta-blocker) prevented hypoglycemia-associated autonomic failure development in rats made recurrently hypoglycemic. Consistent with these findings, propranolol, which crosses blood brain barrier and blocks beta-2 adrenergic receptors, has been shown to prevent hypoglycemia-associated autonomic failure in healthy human subjects. Thus, an intervention which can block the propagating mechanism(s) (i.e. repeated activation of beta2-adrenergic receptors) will likely lead to sympathoadrenal function improvement, and thus increase hypoglycemic symptoms and hypoglycemia awareness.

Beta-blocker is one of the most extensively used medication classes in the United States, and has been commonly utilized in diabetes patients for cardiac diseases. Although beta-blocker may theoretically attenuate hypoglycemic symptoms or lead to worsening of hypoglycemia, multiple studies have proven that beta-blockers increase hypoglycemic symptoms and can be safely used in insulin-dependent diabetes patients. In particular, a retrospective study included more than 13,000 patients and examined the relationship between antihypertensive use and hypoglycemia, and this study supported that beta-blocker use was not associated with an increase in severe hypoglycemia. As well, in a recent post-hoc analysis of a large type 2 diabetes intensive insulin therapy study (ACCORD), the group receiving beta-blocker and intensive insulin therapy had fewer cardiovascular events and comparable all-cause and cardiovascular death events compared to the group receiving beta-blocker and conventional therapy; this is thus evident for the safety of beta-blocker usage in patients undergoing intensive insulin therapy. With the safety data and previous basic/clinical observations, it is therefore proposed that propranolol is a strong testing candidate for potential hypoglycemia-associated autonomic failure treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 1 diabetes mellitus for more than 5 years with impaired awareness of hypoglycemia
* Age between 21 to 59 years old
* Hemoglobin A1c ≤ 9%; most recent value within 3 months
* No beta-blocker use history in the last 6 months
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* History of coronary, cerebral or peripheral vascular disease
* History of cardiac conduction abnormality or heart failure
* History of advanced liver disease
* Active malignancy
* Major Central or Peripheral Nervous System disease
* History of human immunodeficiency virus infection
* Contraindication to beta-blockers, including hypersensitivity to beta-blocker and bronchospastic disease
* Female in pregnancy or not able to practice effective contraception during the study period
* Concomitant acetaminophen use
* Currently utilizing unblinded real-time continuous glucose monitoring
* Advanced diabetic microvascular complications including retinopathy, neuropathy and nephropathy
* Inability to understand or cooperate with study procedure, including performing glucometer glucose assessment a minimum of four times a day, carrying glucose tablets and following standardized hypoglycemia treatment, completing hypoglycemia diary, wearing continuous glucose monitoring, and using a single glucometer
* Recent or current use or involvement in clinical studies of other therapies (e.g. opioid antagonist, SSRI, behavioral modification, relaxation of glycemic control) that may improve hypoglycemia awareness or prevent impaired hypoglycemia awareness development

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anu Sharma, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Hypoglycemia in the Diabetes Control and Complications Trial. The Diabetes Control and Complications Trial Research Group. Diabetes. 1997 Feb;46(2):271-86. PMID 9000705
- [Background] Cryer PE. The barrier of hypoglycemia in diabetes. Diabetes. 2008 Dec;57(12):3169-76. doi: 10.2337/db08-1084. No abstract available. PMID 19033403
- [Background] Cryer PE. Mechanisms of hypoglycemia-associated autonomic failure in diabetes. N Engl J Med. 2013 Jul 25;369(4):362-72. doi: 10.1056/NEJMra1215228. No abstract available. PMID 23883381
- [Background] Geddes J, Schopman JE, Zammitt NN, Frier BM. Prevalence of impaired awareness of hypoglycaemia in adults with Type 1 diabetes. Diabet Med. 2008 Apr;25(4):501-4. doi: 10.1111/j.1464-5491.2008.02413.x. PMID 18387080
- [Background] Cranston I, Lomas J, Maran A, Macdonald I, Amiel SA. Restoration of hypoglycaemia awareness in patients with long-duration insulin-dependent diabetes. Lancet. 1994 Jul 30;344(8918):283-7. doi: 10.1016/s0140-6736(94)91336-6. PMID 7914259
- [Background] Dagogo-Jack S, Rattarasarn C, Cryer PE. Reversal of hypoglycemia unawareness, but not defective glucose counterregulation, in IDDM. Diabetes. 1994 Dec;43(12):1426-34. doi: 10.2337/diab.43.12.1426. PMID 7958494
- [Background] Rickels MR, Peleckis AJ, Markmann E, Dalton-Bakes C, Kong SM, Teff KL, Naji A. Long-Term Improvement in Glucose Control and Counterregulation by Islet Transplantation for Type 1 Diabetes. J Clin Endocrinol Metab. 2016 Nov;101(11):4421-4430. doi: 10.1210/jc.2016-1649. Epub 2016 Aug 29. PMID 27571180
- [Background] Szepietowska B, Zhu W, Chan O, Horblitt A, Dziura J, Sherwin RS. Modulation of beta-adrenergic receptors in the ventromedial hypothalamus influences counterregulatory responses to hypoglycemia. Diabetes. 2011 Dec;60(12):3154-8. doi: 10.2337/db11-0432. Epub 2011 Oct 19. PMID 22013013
- [Background] Chan O, Sherwin R. Influence of VMH fuel sensing on hypoglycemic responses. Trends Endocrinol Metab. 2013 Dec;24(12):616-24. doi: 10.1016/j.tem.2013.08.005. Epub 2013 Sep 21. PMID 24063974
- [Background] Barnes MB, Lawson MA, Beverly JL. Rate of fall in blood glucose and recurrent hypoglycemia affect glucose dynamics and noradrenergic activation in the ventromedial hypothalamus. Am J Physiol Regul Integr Comp Physiol. 2011 Dec;301(6):R1815-20. doi: 10.1152/ajpregu.00171.2011. Epub 2011 Sep 28. PMID 21957162
- [Background] Ramanathan R, Cryer PE. Adrenergic mediation of hypoglycemia-associated autonomic failure. Diabetes. 2011 Feb;60(2):602-6. doi: 10.2337/db10-1374. PMID 21270270
- [Background] UK Prospective Diabetes Study Group. Efficacy of atenolol and captopril in reducing risk of macrovascular and microvascular complications in type 2 diabetes: UKPDS 39. UK Prospective Diabetes Study Group. BMJ. 1998 Sep 12;317(7160):713-20. PMID 9732338
- [Background] Barnett AH, Leslie D, Watkins PJ. Can insulin-treated diabetics be given beta-adrenergic blocking drugs? Br Med J. 1980 Apr 5;280(6219):976-8. doi: 10.1136/bmj.280.6219.976. PMID 6106521
- [Background] Shorr RI, Ray WA, Daugherty JR, Griffin MR. Antihypertensives and the risk of serious hypoglycemia in older persons using insulin or sulfonylureas. JAMA. 1997 Jul 2;278(1):40-3. PMID 9207336
- [Background] Kerr D, MacDonald IA, Heller SR, Tattersall RB. Beta-adrenoceptor blockade and hypoglycaemia. A randomised, double-blind, placebo controlled comparison of metoprolol CR, atenolol and propranolol LA in normal subjects. Br J Clin Pharmacol. 1990 Jun;29(6):685-93. doi: 10.1111/j.1365-2125.1990.tb03689.x. PMID 1974143
- [Background] Viberti GC, Keen H, Bloom SR. Beta blockade and diabetes mellitus: effect of oxprenolol and metoprolol on the metabolic, cardiovascular, and hormonal response to insulin-induced hypoglycemia in normal subjects. Metabolism. 1980 Sep;29(9):866-72. doi: 10.1016/0026-0495(80)90126-2. PMID 6106148
- [Background] Marengo C, Marena S, Renzetti A, Mossino M, Pagano G. Beta-blockers in hypertensive non-insulin-dependent diabetics: comparison between penbutolol and propranolol on metabolic control and response to insulin-induced hypoglycemia. Acta Diabetol Lat. 1988 Apr-Jun;25(2):141-8. doi: 10.1007/BF02581378. PMID 3066086
- [Background] Clausen-Sjobom N, Lins PE, Adamson U, Curstedt T, Hamberger B. Effects of metoprolol on the counter-regulation and recognition of prolonged hypoglycemia in insulin-dependent diabetics. Acta Med Scand. 1987;222(1):57-63. doi: 10.1111/j.0954-6820.1987.tb09929.x. PMID 3307308
- [Background] Odugbesan O, Toop M, Barnett AH. Beta-and alpha-adrenergic blockade and metabolic responses to insulin induced hypoglycaemia in diabetics. Diabetes Res. 1987 Jul;5(3):135-8. PMID 2822334

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propranolol | Placebo
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Self-reported Hypoglycemic Episodes to Total Hypoglycemic Episodes Determined by Continuous Glucose Monitoring (CGM)
Description: A subject's self-reported hypoglycemic episode is defined by a hypoglycemic symptom record on the hypoglycemia diary with a confirmatory glucose value (glucometer value < 70 mg/dL), or an incidental glucometer value < 70 mg/dL if no hypoglycemia symptom develops. A single CGM hypoglycemic episode is defined by any CGM readings < 70 mg/dL, followed by at least one reading ≥ 70 mg/dL from the Dexcom Professional Mobile CGM system. Self-reported and CGM assessment of hypoglycemic episodes will be conducted for two weeks before study drug intervention and two weeks after study drug intervention. The average change in the ratio of self-reported hypoglycemic episodes to total (CGM) episodes will be compared between the propranolol and placebo treatment arms
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Gold Questionnaire Score for Hypoglycemia Awareness
Description: Subjects will complete the Gold questionnaire for hypoglycemia awareness at the baseline and at the last visit of the intervention period. The Gold questionnaire is comprised of one question to evaluate the hypoglycemia awareness, with scores from 1 to 7, representing from normal to minimal/no hypoglycemia awareness. The average change in Gold questionnaire score from baseline to the last visit will be compared between the propranolol and placebo treatment arms.
Time Frame: 4 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Clarke Questionnaire Score for Hypoglycemia Awareness
Description: Subjects will complete the Clarke questionnaire for hypoglycemia awareness at the baseline and at the last visit of the intervention period. The Clarke questionnaire is comprised of eight questions to evaluate the hypoglycemia awareness. The answer for each individual question will represent a score (0 or 1). These scores will be summed together to a final score from 0 to 7, representing from normal to minimal/no hypoglycemia awareness. The average change in Clarke questionnaire score from baseline to the last visit will be compared between the propranolol and placebo treatment arms.
Time Frame: 4 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pederson-Bjergaard Questionnaire Score for Hypoglycemia Awareness
Description: Subjects will complete the Pederson-Bjergaard questionnaire for hypoglycemia awareness at the baseline and at the last visit of the intervention period. The Pederson-Bjergaard questionnaire is comprised of one question to evaluate the hypoglycemia awareness, with answers of "Always", "sometimes", "occasionally", "never" or "Do not know". Each answer will represent an awareness status. The change in Pederson-Bjergaard questionnaire status from baseline to the last visit will be compared between the propranolol and placebo treatment arms.
Time Frame: 4 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Nadir Glucose Level
Description: Nadir glucose level during each hypoglycemic episode will be detected by CGM during a 2-week interval at baseline and at the end of the treatment period. The average of nadir blood glucose levels will be calculated and the change will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Nadir Glucose Level in Categories
Description: Nadir glucose level during each hypoglycemic episode will be detected by CGM during a 2-week interval at baseline and at the end of the treatment period. The number of hypoglycemic events will be totaled in the severity categories of nadir glucose level: < 70 mg/dL; < 60 mg/dL; < 56 mg/dL; < 50 mg/dL; and < 40 mg/dL. The change in the number of hypoglycemic events in these categories will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Hypoglycemia Duration
Description: Duration of hypoglycemia will be detected by CGM during a 2-week interval at baseline and at the end of the treatment period. The total duration of hypoglycemia (in minutes) will be calculated for each duration categories of hypoglycemia: <15 minutes, ≥ 15 minutes, ≥ 30 minutes, ≥ 45 minutes and ≥ 60 minutes. The change in the total time of hypoglycemia in these categories will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Blood Glucose Area Under the Curve (AUC)
Description: Blood glucose will be detected by CGM during a 2-week interval at baseline and at the end of the treatment period. The AUC of blood glucose will be calculated for each severity categories of nadir glucose level: < 70 mg/dL; < 60 mg/dL; < 56 mg/dL; < 50 mg/dL; and < 40 mg/dL. The change in AUC of these categories will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Duration of Hypoglycemia Onset-to-Diagnosis
Description: The time of hypoglycemic symptom and glucometer reading of each hypoglycemic episode will be documented by study subjects in the hypoglycemia diary, and the onset time of hypoglycemia will be detected by CGM during a 2-week interval at baseline and at the end of the treatment period. The duration of hypoglycemia onset-to-diagnosis will be calculated as the time difference between hypoglycemia onset as recorded on CGM, and documented hypoglycemic symptom and glucometer reading, whichever is the earliest. The change in the average duration of hypoglycemia onset-to-diagnosis will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Duration of Hypoglycemia Onset-to-Treatment
Description: The time of hypoglycemia treatment of each hypoglycemic episode will be documented by study subjects in the hypoglycemia diary, and the onset time of hypoglycemia will be detected by CGM during a 2-week interval at baseline and at the end of the treatment period. The duration of hypoglycemia onset-to-treatment will be calculated as the time difference between hypoglycemia onset as recorded on CGM, and documented hypoglycemia treatment. The change in the average duration of hypoglycemia onset-to-treatment will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Duration of Hypoglycemia Diagnosis-to-Recovery
Description: The time of hypoglycemic symptom and glucometer reading of each hypoglycemic episode will be documented by study subjects in the hypoglycemia diary, and the recovery time of hypoglycemia will be detected by CGM during a 2-week interval at baseline and at the end of the treatment period. The duration of hypoglycemia diagnosis-to-recovery will be calculated as the time difference between the documented hypoglycemic symptom and glucometer reading, whichever is the earliest, and hypoglycemia recovery as recorded on CGM. The change in the average duration of hypoglycemia diagnosis-to-recovery will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Duration of Hypoglycemia Treatment-to-Recovery
Description: The time of hypoglycemia treatment of each hypoglycemic episode will be documented by study subjects in the hypoglycemia diary, and the recovery time of hypoglycemia will be detected by CGM during a 2-week interval at baseline and at the end of the treatment period. The duration of hypoglycemia treatment-to-recovery will be calculated as the time difference between the documented hypoglycemia treatment and hypoglycemia recovery as recorded on CGM. The change in the average duration of hypoglycemia treatment-to-recovery will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Total Hypoglycemia Episodes
Description: Hypoglycemia will be reported by patients detected by CGM during a 2-week interval at the baseline and at end of the treatment period. The total number of hypoglycemic episodes as defined by CGM readings of < 70 mg/dL will be counted, and the changes in the number will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Total Severe Hypoglycemia Episodes
Description: Severe hypoglycemia is a clinical event defined by any hypoglycemic episode requiring outside help in the treatment administration of the particular hypoglycemic episode. Severe hypoglycemia episodes will be recorded by hypoglycemia diary during a 2-week interval at baseline and at the end of the treatment period. The total number of hypoglycemia/severe hypoglycemia episodes as defined by CGM readings of < 70 mg/dL will be counted and the change will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 week
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Fear of Hypoglycemia Score
Description: Subjects will complete the Fear of Hypoglycemia Questionnaire at baseline and the last visit of the intervention period. The average change in Fear of Hypoglycemia Questionnaire score from baseline to 4 weeks will be compared between the propranolol and placebo treatment arms.
Time Frame: 4 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Mean Blood Glucose
Description: Blood glucose will be detected by CGM during a 2-week interval at the baseline and at the end of the treatment period. The average change will be compared between the propranolol and placebo treatment arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Propranolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT03161964/Prot_SAP_000.pdf